CLINICAL TRIAL: NCT06528990
Title: Perioperative Ostomy Self-Management Telehealth Intervention for Cancer Survivors
Brief Title: Telehealth Intervention for Ostomy Self-Management
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: City of Hope Medical Center (Other)
Collaborators: United States Department of Defense (U.S. Federal Agency)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: 24275
Record Dates: First submitted 2024-07-26; First posted 2024-07-31 (Actual); Last update posted 2025-02-25 (Actual); Status verified 2025-02

CONDITIONS: Colorectal Cancer; Bladder Cancer
Keywords: Ostomy, colorectal cancer, bladder cancer, quality of liffffffffffffffffffffe, telehealth, family caregivers
MeSH Terms: conditions — Colorectal Neoplasms; Urinary Bladder Neoplasms | interventions — Standard of Care

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Periop-OSMT Telehealth Intervention Arm (Experimental): Arm 1 includes the following key components: 1) assignment to a peer ostomate; 2) ostomy self-management skills building delivered through group telehealth sessions and led by trained ostomy nurses and peer ostomates; 3) intervention resource manual. The intervention is delivered through 2 telephone and 5 telehealth sessions over a 16 week period.
  Interventions: Behavioral: Telehealth Intervention
- Standard of Care Arm (Other): Arm 2 involves standard of care, where patients and family caregivers are managed by the oncology care team. Care may include clinic visits for follow-up, cancer directed treatments, referrals to other medical specialties as needed, and institutional ostomy nurse support before and after surgery as needed.
  Interventions: Other: Standard of care

INTERVENTIONS:
Behavioral: Telehealth Intervention — This includes the following key components: 1) assignment to a peer ostomate; 2) ostomy self-management skills building delivered through group telehealth sessions and led by trained ostomy nurses and peer ostomates; 3) intervention resource manual.
  Arms: Periop-OSMT Telehealth Intervention Arm
Other: Standard of care — standard of care, where patients and family caregivers are managed by the oncology care team. Care may include clinic visits for follow-up, cancer directed treatments, referrals to other medical specialties as needed, and institutional ostomy nurse support before and after surgery as needed.
  Arms: Standard of Care Arm

SUMMARY:
Over one million individuals in the U.S. have ostomies. An ostomy is a surgical procedure that creates an opening in the abdominal wall that allows bodily waste (urinary or fecal) to pass through into an external pouch; in essence, it is the externalization of the gastrointestinal or urinary structures to the abdominal wall. For cancer, ostomies are most commonly placed for rectal cancers, followed by urinary bladder cancer. The health-related quality of life impact of an ostomy is tremendous and greater than many other cancer treatments. The goal of this study is to pilot-test a perioperative ostomy self-management telehealth intervention (Periop-OSMT) in patients with colorectal and bladder cancer and their family caregivers. Participants will receive seven group telehealth sessions before and after ostomy surgery. This pilot clinical trial will study the feasibility of the methods/interventions and determine the preliminary efficacy to support a larger confirmatory trial.

DETAILED DESCRIPTION:
An ostomy is a disability that adversely affects the HRQOL of cancer survivors and their support persons/family caregivers (FCGs) at all phases of cancer survivorship. More than half of survivors experience stoma-related challenges such as pain, troublesome odor, skin problems around the stoma, and leakage. Ongoing problems include pouching care, travel out of the home (especially relevant for rural populations), social interactions, intimacy, and acceptance of/satisfaction with appearance. Studies document persistent challenges including sexuality, psychological problems, and interference with work, and recreation and sporting activities. The purpose of this study is to assess the feasibility of a perioperative ostomy self-management telehealth intervention (Periop-OSMT) and to determine the preliminary efficacy of the intervention on participant-reported outcomes, compared to the usual care arm. We hypothesize that the intervention will be feasible, acceptable and will demonstrate preliminary improvements in outcomes compared to the usual care arm.

ELIGIBILITY:
Patient Eligibility Criteria:

* Patient with bladder or colorectal cancer
* Scheduled to undergo a surgical procedure that includes the creation of an intestinal stoma (fecal or urinary, permanent or temporary)
* For bladder cancer, only patients with incontinent urostomies (ileal conduit) are eligible.
* Age: ≥ 18 years
* Ability to read and understand English for Questionnaires

Family Caregiver Eligibility Criteria:

* A family member or friend identified by the patient and defined as a person who knows the patient well and is involved in the patient's care before and after surgery
* Age: ≥ 18 years
* Ability to read and understand English for Questionnaires
* Pregnant FCGs are eligible for participation. Participation in this behavioral/educational intervention should not impact the pregnancy/fetus.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 150 (Estimated)
Dates: Start 2025-01-02 (Actual); Primary Completion 2028-06-04 (Estimated); Study Completion 2028-06-04 (Estimated)

PRIMARY OUTCOMES:
Self-Efficacy for Ostomy Self-Management | At 13 weeks post-randomization
  Will be measured by the Self-Efficacy to Perform Self-management Behaviors Scale, an outcome measure for Chronic Disease Management Interventions, this scale represents 8 domains: physical activity, information seeking, support, communication with HC providers, ostomy management, social and recreational, symptom management, and depression. Higher scores reflect better self-efficacy. Study arm differences at 13 weeks will be assessed via repeated measures linear regression models with adjustment for baseline value of the outcome and stratification factors including cancer type (bladder versus colorectal) and whether the patient has a caregiver.

OTHER OUTCOMES:
Feasibility of the Intervention | at baseline, 13 weeks, 26 weeks post randomization
  Will be measured by a) at least 60% of eligible participants enrolled, b) at least 60% of participants completing at least ≥80% of the intervention (at least one of sessions 1-2 and all of sessions 3-6), c) at least 60% of participants that complete any follow-up assessments after randomization, and d) exploring participant experience with the intervention through structured exit interviews).
Patient Activation | At 13 and 26 weeks post-randomization
  Will be measured by the Patient Activation Measure (PAM). The measure assessed four stages: (1) believing the patient role is important, (2) having the confidence and knowledge necessary to take action, (3) actually taking action to maintain and improve one's health, and (4) staying the course even under stress. Higher scores reflect higher activation. Study arm differences at 13 weeks and 26 weeks will be assessed via repeated measures linear regression models with adjustment for baseline value of the outcome and stratification factors including cancer type (bladder versus colorectal) and whether the patient has a caregiver.
Patient and Family Caregiver Psychological Distress | At Baseline, 13 and 26 weeks post-randomization
  Will be measured by the Distress Thermometer. The tool evaluates psychological distress over the past week, based on a scale of 0 (no distress) to 10 (extremely distressed). A cut-off of 3/10 indicates a need for intervention. Study arm differences at 13 weeks and 26 weeks will be assessed via repeated measures linear regression models with adjustment for baseline value of the outcome and stratification factors including cancer type (bladder versus colorectal) and whether the patient has a caregiver.
Quality of Life | At Baseline, 13 and 26 weeks post-randomization
  Will be measured by the City of Hope-Quality of Life-Colorectal Cancer (COH-QOL-CRC). Evaluates overall HRQOL and four dimensions: physical, psychological, social, and spiritual well-being. Higher score reflect better quality of life. Study arm differences at 13 weeks and 26 weeks will be assessed via repeated measures linear regression models with adjustment for baseline value of the outcome and stratification factors including cancer type (bladder versus colorectal) and whether the patient has a caregiver.
Family Caregiver Quality of Life | At Baseline, 13 and 26 weeks post-randomization
  Will be measured by the City of Hope-Quality of Life-Family (COH-QOL-Family) tool. Measures the FCG QOL in the physical, psychological, social, and spiritual well-being domains. Ordinal scale ranges from 0-10, with higher scores indicating better QOL. Study arm differences at 13 weeks and 26 weeks will be assessed via repeated measures linear regression models with adjustment for baseline value of the outcome and stratification factors including cancer type (bladder versus colorectal) and whether the patient has a caregiver.
Colostomy Impact | At Baseline, 13 and 26 weeks post-randomization
  Will be measured by the Colostomy Impact Score and used in patients with colorectal cancer only. Identifies patients with stoma dysfunction that impairs HRQOL by dividing patients into 'minor' and 'major' CI groups.

CONTACTS AND LOCATIONS:
Overall Officials: Virginia Sun, PhD, RN, Principal Investigator — City of Hope Medical Center
Locations (1):
- City of hope Medical Center, Duarte, California, United States